CLINICAL TRIAL: NCT06072053
Title: YL-1 Needle Puncture Versus Burr-hole Craniotomy With Postoperative Exhaustive Drainage for Chronic Subdural Hematoma: a Multicenter Prospective Cohort Study
Brief Title: YL-1 Needle Puncture vs BHC With Postoperative Exhaustive Drainage for CSDH
Acronym: NEBULA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Weiming Liu, Professor, Beijing Tiantan Hospital
Other Study IDs: HX-B-2023035
Record Dates: First submitted 2023-10-01; First posted 2023-10-10 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic Subdural Hematoma; YL-1 Needle Drainage; Burr Hole Craniostomy; Exhaustive drainage strategy
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BHC group: Patients with CSDH recruited from the neurosurgery departments of 6 medical centers in China who had clinically significant symptoms confirmed by computed tomography or magnetic resonance imaging and ultimately treated with Bulr-hole Craniotomy.
  Interventions: Procedure: Burr Hole Craniostomy and Postoperative Exhaustive Drainage Strategy
- YL-1 Needle Puncture group: Patients with CSDH recruited from the neurosurgery departments of 6 medical centers in China who had clinically significant symptoms confirmed by computed tomography or magnetic resonance imaging and ultimately treated with YL-1 needle puncture.
  Interventions: Procedure: YL-1 puncture needle and Postoperative Exhaustive Drainage Strategy

INTERVENTIONS:
Procedure: Burr Hole Craniostomy and Postoperative Exhaustive Drainage Strategy — According to the preoperative CT results, drilling and drainage was performed at the thickest level of the hematoma; during the operation, the hematoma cavity was adequately flushed with saline and a drainage tube was left in the hematoma cavity; after the operation, the hematoma cavity was flushed with urokinase, and the drainage tube was removed after adequate drainage.
  Groups: BHC group
Procedure: YL-1 puncture needle and Postoperative Exhaustive Drainage Strategy — Based on preoperative CT, the thickest level of the hematoma was selected and localized. During the operation, an electric drilling needle was used to rapidly break through the skull and dura to enter the cavity of the subdural hematoma, and the puncture needle was fixed to the skull to drain the subdural hematoma. After the operation, the hematoma cavity was flushed with urokinase, and the drainage tube was removed after adequate drainage.
  Groups: YL-1 Needle Puncture group

SUMMARY:
A prospective multicenter cohort study was designed to compare the differences in complications with YL-1 Needle Puncture versus Bulr-hole Craniotomy (BHC) with postoperative Exhaustive Drainage strategy for patients with Chronic Subdural Hematoma.

DETAILED DESCRIPTION:
Chronic subdural haematoma (CSDH) is a common condition in neurosurgery. It is generally considered to be a closed exudate formed by blood or blood degradation products between the dura mater and the arachnoid membrane. Its local occupying effect will compress the neighbouring brain tissues, leading to varying degrees of neurological dysfunction. In severe cases, it can lead to cerebral hernia and endanger the patient's life. Currently, the most commonly used surgical method for the treatment of chronic subdural haematoma is BHC, but many studies have found that various complications may occur after BHC. With the rapid development of neurosurgical microtechnology, Twist Drill Craniotomy (TDC) was proposed. YL-1 puncture needle technique, as a modified solution of TDC, has a short surgical time and is less traumatic to patients. In the treatment of chronic subdural haematomas, investigator's team has adopted the strategy of postoperative instillation of urokinase and adequate drainage of the haematoma. Based on this, this study intends to conduct a multicentre prospective observational cohort study of the above two treatment in order to scientifically and rigorously derive the optimal clinical treatment strategy for chronic subdural haematoma.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, male or female, 18 years ≤ age ≤ 90 years;
2. Preoperative neurological dysfunction, such as headache and dizziness, nausea and vomiting, limb numbness or weakness, unsteady walking, limb twitching, confusion, aphasia, slow response, memory loss, etc;
3. A definite diagnosis of chronic subdural hematoma by CT or MRI;
4. Signed informed consent.

Exclusion Criteria:

1. No symptoms before surgery and no obvious impact on oneself's normal life;
2. Lack of mass effect, less than 0.5 cm of midline structure shift, and no need surgery judged clinically by neurosurgeons;
3. Previous surgery for chronic subdural hematoma during the past 6 months;
4. Previous intracranial surgery for any neurological disorders but chronic subdural hematoma before
5. Existing poor medication condition or severe comorbidity so that surgery cannot be tolerated or follow-up cannot be completed
6. Combination of major systemic diseases that are expected to interfere with study implementation and follow-up observations;
7. Definite coagulation abnormalities with a high risk of bleeding (presence of one of the following three: prolongation of the prothrombin time PT or the activated partial thromboplastin time APTT by more than 10 seconds, an international normalized ratio INR greater than 3.0, and an absolute platelet value of less than 100 × 109/L);
8. Postoperative cooperation is suspected to be insufficient for follow-up for 6 months;
9. Reproductive-age women without verified negative pregnancy testing;
10. Participating in other research

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with CSDH recruited from the neurosurgery departments of 12 medical centers in China who had significant clinical symptoms confirmed by computed tomography or magnetic resonance imaging. Six medical centers each used BHC as well as YL-1 puncture needles for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Complication rates | From operation up to 3 months postoperatively
  To compare the difference in overall complication rates between the two groups of CSDH patients treated with YL-1 perforator needles and drilled drainage at 3 months postoperatively.

SECONDARY OUTCOMES:
Recurrence rate | From operation up to 3 months postoperatively
  To compare the difference in recurrence rate at 3 months postoperatively between the two groups;
Mortality rate | From operation up to 3 months postoperatively
  To compare the difference in mortality rate at 3 months postoperatively between the two groups;
Change of Modified Rankin Scale (MRS) between groups from baseline to 3 months after operation | At baseline and at 3 months after operation
  Modified Rankin Scale ranges from score 1 to 6, and higher scores mean a worse clinical outcome, where score 1 indicates normal daily functionality and score 6 indicates death.
Quality of life assessment (EQ-5D-5L) | At baseline and at 3 months after operation
  A standardized instrument, EuroQoL 5-Dimension 5-Level (EQ-5D-5L) questionnaire, will be used as a generic measure of health related quality of life. The questionnaire contains 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension rates across five levels, including 'No problems-Slight problems-Moderate problems-Severe problems-Unable to'postoperatively between the two groups.
Change of Markwalder Grading Scale between groups from baseline to 3 months after operation | At baseline and at 3 months after operation
  Markwalder Grading Scale ranges from grade 0 to 4, and higher scores mean a worse neurological outcome, where grade 0 indicates normal neurological function and grade 4 indicates coma.
Hospitalization costs | At baseline.
  To compare the difference in hospitalization costs between the two groups.
Length of hospitalization | At baseline.
  To compare the difference in length of hospitalization between the two groups;

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Liu, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almenawer SA, Farrokhyar F, Hong C, Alhazzani W, Manoranjan B, Yarascavitch B, Arjmand P, Baronia B, Reddy K, Murty N, Singh S. Chronic subdural hematoma management: a systematic review and meta-analysis of 34,829 patients. Ann Surg. 2014 Mar;259(3):449-57. doi: 10.1097/SLA.0000000000000255. PMID 24096761
- [Background] Brennan PM, Kolias AG, Joannides AJ, Shapey J, Marcus HJ, Gregson BA, Grover PJ, Hutchinson PJ, Coulter IC; British Neurosurgical Trainee Research Collaborative. The management and outcome for patients with chronic subdural hematoma: a prospective, multicenter, observational cohort study in the United Kingdom. J Neurosurg. 2017 Mar 17:1-8. doi: 10.3171/2016.8.JNS16134.test. Online ahead of print. PMID 28306417
- [Background] Duerinck J, Van Der Veken J, Schuind S, Van Calenbergh F, van Loon J, Du Four S, Debacker S, Costa E, Raftopoulos C, De Witte O, Cools W, Buyl R, Van Velthoven V, D'Haens J, Bruneau M. Randomized Trial Comparing Burr Hole Craniostomy, Minicraniotomy, and Twist Drill Craniostomy for Treatment of Chronic Subdural Hematoma. Neurosurgery. 2022 Aug 1;91(2):304-311. doi: 10.1227/neu.0000000000001997. Epub 2022 May 24. PMID 35593710
- [Background] Kolias AG, Chari A, Santarius T, Hutchinson PJ. Chronic subdural haematoma: modern management and emerging therapies. Nat Rev Neurol. 2014 Oct;10(10):570-8. doi: 10.1038/nrneurol.2014.163. Epub 2014 Sep 16. PMID 25224156
- [Background] Lee SJ, Hwang SC, Im SB. Twist-Drill or Burr Hole Craniostomy for Draining Chronic Subdural Hematomas: How to Choose It for Chronic Subdural Hematoma Drainage. Korean J Neurotrauma. 2016 Oct;12(2):107-111. doi: 10.13004/kjnt.2016.12.2.107. Epub 2016 Oct 31. PMID 27857917